CLINICAL TRIAL: NCT04202380
Title: Different Azithromycin Protocols for Management of Preterm Pre-labor Rupture of Membranes
Brief Title: Azithromycin for Preterm Pre-labor Rupture of Membranes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A-PROM
Record Dates: First submitted 2019-12-16; First posted 2019-12-17 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Preterm Pre-labor Rupture of Membranes
MeSH Terms: interventions — Azithromycin; Ampicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Azithromycin 1 day group (Other): Patients will receive Azithromycin 1000mg once orally
  Interventions: Drug: Azithromycin; Drug: Ampicillin
- Azithromycin 5 days group (Other): Patients will receive Azithromycin 500mg once orally, followed by Azithromycin 250mg orally daily for 4 days
  Interventions: Drug: Azithromycin; Drug: Ampicillin

INTERVENTIONS:
Drug: Azithromycin — Patients will receive Azithromycin orally 1000 mg
Drug: Ampicillin — All patients will receive Ampicillin 2gm IV every 6 hours for 2 days
Drug: Azithromycin — Azithromycin 500 mg orally once
  Arms: Azithromycin 5 days group
Drug: Azithromycin — Azithromycin 250 mg orally daily for 4 days
  Arms: Azithromycin 5 days group

SUMMARY:
The preterm prelabour rupture of membranes is defined as the spontaneous rupture of the fetal membranes before 37 completed weeks. Preterm prelabour rupture of membranes complicates up to 3% of pregnancies and is associated with 30-40% of preterm births. preterm prelabour rupture of membranes can result in significant neonatal morbidity and mortality, primarily from prematurity, sepsis, cord prolapse, and pulmonary hypoplasia. In addition, there are risks associated with chorioamnionitis and placental abruption The diagnosis of spontaneous rupture of the membranes is made by maternal history followed by a sterile speculum examination. If on speculum examination, no amniotic fluid is observed, clinicians should consider performing an insulin-like growth factor-binding protein-1 or placental alpha microglobulin-1 test of vaginal fluid to guide further management.

One of the risks associated with preterm prelabour rupture of membranes is ascending infection leading to chorioamnionitis, and subsequent fetal and neonatal infection.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age is between 28 wks and 37wks
2. Singleton living pregnancy.
3. Confirmed Premature Pre-labor rupture of membranes (PPROM).

Exclusion Criteria:

1. previable rupture of membranes (<23+6wks)
2. Multiple gestations
3. Macrolide allergy
4. patient receiving combination macrolide therapy
5. lethal fetal anomalies
6. contraindications to expectant management of PPROM at time of diagnosis e.g. concurrent preterm labor, placental abruption, chorioamnionitis or non-reassuring fetal testing

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Days from diagnosis of preterm pre-labor rupture of membranes to delivery. | 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital - Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Abdelfattah LE, Aboshama RA, Abdelbadie AS, Abulhasan MH, Anan MA, Abdelaal II. Different azithromycin protocols for management of preterm prelabour rupture of membranes: a randomized clinical trial. BMC Pregnancy Childbirth. 2022 Nov 23;22(1):869. doi: 10.1186/s12884-022-05189-7. PMID 36424542